CLINICAL TRIAL: NCT06876181
Title: In Vivo Study of Local Tranexamic Acid Concentrations Following Intra-Articular Administration in Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Valdoltra Orthopedic Hospital (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: J3-3067; J3-3067 (Other Grant/Funding Number: Slovenian Research Agency (ARRS))
Record Dates: First submitted 2025-03-09; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Local Concentration of Tranexamic Acid Following Intra-articular Administration in TKA
Keywords: Tranexamic acid; Intra-articular administration; topical administration; Local concentration; Elimination half-time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of postoperative periarticular haematoma obtained via a drainage catheter inserted into the knee joint space.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Recruited subjects with end-stage knee joint osteoarthritis
  Interventions: Other: Pharmacokinetics of Intra-Articularly Administered TXA: Postoperative Concentration Dynamics in Periarticular Hematoma

INTERVENTIONS:
Other: Pharmacokinetics of Intra-Articularly Administered TXA: Postoperative Concentration Dynamics in Periarticular Hematoma — As part of the standard total knee arthroplasty procedure, participants receive a 2 g dose of tranexamic acid into the joint space after suturing the joint capsule. Before closing the joint capsule, a silicone drain is inserted into the joint space, through which periarticular hematoma samples are collected aseptically at 0.5, 1.5, 3, 6, and 9 hours post-application.

SUMMARY:
The goal of this observational study is to measure local tranexamic acid (TXA) concentrations following intra-articular administration in patients undergoing total knee arthroplasty. By evaluating its pharmacokinetic profile in the periarticular hematoma, the study will also assess the safety of topically administered TXA considering its cytotoxicity in healthy periarticular tissue. The main questions it aims to answer are:

* How does TXA concentration in periarticular hematoma change over time following intra-articular administration after TKA?
* Do local TXA concentrations after standard intra-articular dose of 2 g exceed the proposed cytotoxic levels, and for how long?

Participants will:

* Receive standard 2 g of TXA intra-articularly at the end of surgery as per the estabished hospital protocol
* Undergo intra-articular hematoma fluid sampling via a drainage catheter at 0.5, 1.5, 3, 6, and 9 hours postoperatively

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of advanced osteoarthritis of the knee joint

Exclusion Criteria:

* known allergy to TXA
* family history or past spontaneous thromboembolic event
* pathological preoperative blood analysis
* advanced heart failure (NYHA > 2)
* ischemic heart disease
* epilepsy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from Valdoltra Orthopaedic Hospital between August 2022 and March 2023.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Tranexamic acid concentrations in periarticular hematoma at 0.5, 1.5, 3, 6, and 9 hours following a standard intra-articular injection of 2 g of tranexamic acid | From the collection of samples after the total knee arthroplasty procedure to the analysis of hematoma samples within 2-3 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Valdoltra Orthopaedic Hospital, Ankaran, Ajdovščina Municipality, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Time Frame: Begining 3 months and ending 1 year after the publication of results.